CLINICAL TRIAL: NCT02958449
Title: Prospective Clinical Investigation for a Randomized, Controlled, Multicenter Non-inferiority Study Comparing Standard Wound Closure Technique With Drains (Control) to Standard Wound Closure Techniques With TissuGlu® and No Drains (Test) in Mastectomy
Brief Title: Prospective Clinical Investigation Comparing Standard Wound Closure Technique With Drains (Control) to Standard Wound Closure Techniques With TissuGlu® and No Drains (Test) in Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cohera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-100-0145
Record Dates: First submitted 2016-11-03; First posted 2016-11-08 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Cancer, Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test - Standard Closure with TissuGlu Surgical Adhesive (Experimental): Standard closure plus treatment with TissuGlu
  Interventions: Device: Test - Standard Closure with TissuGlu Surgical Adhesive
- Control - Standard Closure (No Intervention): Standard closure with no intervention

INTERVENTIONS:
Device: Test - Standard Closure with TissuGlu Surgical Adhesive — Patients randomized into the Test group, TissuGlu® will be applied to the chest wall after removal of the breast tissue using the custom applicator during a standard mastectomy procedure followed by normal wound closure (suturing technique) without drain placement.
  Arms: Test - Standard Closure with TissuGlu Surgical Adhesive

SUMMARY:
Comparing standard wound closure technique with drains (control) to standard wound closure techniques with TissuGlu® and no drains (test) in mastectomy

DETAILED DESCRIPTION:
A prospective, randomized, controlled, multicenter non-inferiority study comparing standard wound closure technique with drains (control) to standard wound closure techniques with TissuGlu® and no drains (test) in mastectomy. Patients will be enrolled for 90 Days from day of Surgery. It is expected that it will take 6-9 months for the full duration of the study including the 90 day follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age;
2. Provide signed and dated informed consent form;
3. Willing to comply with all study procedures, schedules and be available for the follow-up evaluations for the duration of the study;
4. Willing to follow instructions for incision care and follow guidelines related to resumption of daily activities;
5. Agree not to schedule any additional elective surgical procedures that involve an incision until their participation in this study is complete;
6. In good general health in the opinion of the Investigator with no conditions that would significantly impact wound healing as determined by medical history, and review of recent concomitant medications;
7. Requiring a mastectomy (standard, modified, modified radical) with or without sentinel node biopsy;
8. ≤ ASA 3 - American Society of Anesthesiologists Physical Classification System

Exclusion Criteria:

1. Pregnancy or lactation;
2. Known medical condition that results in compromised blood supply to tissues;
3. Known or suspected allergy or sensitivity to any test materials or reagents;
4. Any condition known to affect wound healing, such as collagen vascular disease;
5. Receiving antibiotic therapy for pre-existing condition or infection;
6. Planned immediate breast reconstruction;
7. Concurrent use of fibrin sealants or other internal wound care devices;
8. Unable to understand questions, instructions or the informed consent presentation in the language of the investigators performing the study;
9. Requiring a mastectomy with ALND (as determined at time of surgery);
10. Be participating in any conflicting medical device clinical trial within 30 days of enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-12; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of Post-Operative Clinical Interventions | from day 0 to day 90
  Clinical Intervention is defined as one of the following events:
  1. Removal of an in-dwelling drain (As defined in the Protocol);
  2. Needle aspiration to remove fluid from a Clinically-Relevant Seroma (As defined in the Protocol);
  3. Invasive action to the drain or drain wound such as repositioning or re-attaching the drain retention sutures;
  4. Reinsertion or insertion of a drain post operatively;
  5. Surgical procedures due to wound healing complications related to wound management

SECONDARY OUTCOMES:
Wound healing related complications | Day 1, 5, 14, 30, 90
Cumulative drain volume, aspiration volume, and total wound drainage (drain volume + aspiration volume) | Day 1, 5, 14, 30, 90
Days to drain removal | Day 1, 5, 14, 30, 90
Cumulative days of treatment (with drains or aspiration) | Day 1, 5, 14, 30, 90
Days to discharge from hospital | Day 1, 5, 14, 30, 90
Number of Clinically Relevant Seromas formation (number and aspiration volume) | Day 1, 5, 14, 30, 90
Incidence and timing of initiation of adjuvant therapy related to the mastectomy procedure (such as radiation therapy, chemotherapy, endocrine therapy) | Day 1, 5, 14, 30, 90
Patient Benefit Questionnaire | Day 1, 5, 14, 30, 90

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (4):
  - University Hospital Cologne Holweide, Cologne
  - University Hospital Cologne St. Elisabeth, Cologne
  - University Hospital Erlangen, Erlangen
  - University Hospital Greifswald, Greifswald
- United Kingdom (6):
  - Royal Cornwall Hospital, Cornwall
  - Derby Teaching Hospitals NHS Foundation Trust, Derby
  - University Hospitals of Leicester NHS Foundation Trust, Leicester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Hallamshire Hospital, Sheffield
  - St. Helens & Knowsley Teaching Hospitals NHS Trust, St Helens